CLINICAL TRIAL: NCT02668653
Title: A Phase 3, Double-Blind, Placebo-controlled Study of Quizartinib Administered in Combination With Induction and Consolidation Chemotherapy, and Administered as Continuation Therapy in Subjects 18 to 75 Years Old With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia (QuANTUM First)
Brief Title: Quizartinib With Standard of Care Chemotherapy and as Continuation Therapy in Patients With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia (AML)
Acronym: QuANTUM-First
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC220-A-U302; 2015-004856-24 (EudraCT Number); 173667 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia; Leukemia
Keywords: Newly diagnosed Acute Myeloid Leukemia; FLT3-ITD positive; Chemotherapy; Induction chemotherapy; Consolidation chemotherapy; Quizartinib; Feline McDonough sarcoma (FMS)-like tyrosine kinase 3; AC220; FLT3-ITD; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Drug Therapy; Cytarabine; Daunorubicin; Idarubicin; quizartinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy plus quizartinib (Experimental): Induction: up to 2 cycles with cytarabine and daunorubicin/idarubicin, followed by the experimental drug quizartinib
  Consolidation: up to 4 cycles of cytarabine followed by the experimental drug quizartinib and/or hematopoeitic stem cell transplant
  Continuation: up to 36 cycles with the experimental drug quizartinib
  Interventions: Drug: Chemotherapy; Drug: Quizartinib
- Chemotherapy plus placebo (Active Comparator): Induction: up to 2 cycles with cytarabine and daunorubicin/idarubicin, followed by placebo
  Consolidation: up to 4 cycles of cytarabine followed by placebo and/or hematopoeitic stem cell transplant
  Continuation: up to 36 cycles with placebo
  Interventions: Drug: Chemotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Chemotherapy
  Other Names: Cytarabine; Daunorubicin; Idarubicin
Drug: Quizartinib
  Other Names: Test Product
  Arms: Chemotherapy plus quizartinib
Drug: Placebo
  Other Names: Placebo Control
  Arms: Chemotherapy plus placebo

SUMMARY:
Quizartinib is an experimental drug. It is not approved for regular use. It can only be used in medical research.

Adults might be able to join this study after bone marrow tests show they have a certain kind of blood cancer (FLT3-ITD AML).

Participants will have an equal chance of receiving quizartinib or placebo along with their chemotherapy.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-control global study. The purpose of this study is to compare the effect of quizartinib versus placebo (administered with standard induction and consolidation chemotherapy, then administered as continuation therapy for up to 36 cycles) on overall survival in subjects with FLT3-internal tandem duplication (ITD) positive AML.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date an Ethics Committee (EC) or Institutional Review Board approved Informed Consent Form (ICF) before performance of any study-specific procedures or tests;
2. Is ≥18 years or the minimum legal adult age (whichever is greater) and ≤75 years (at Screening);
3. Newly diagnosed, morphologically documented primary AML or AML secondary to myelodysplastic syndrome or a myeloproliferative neoplasm, based on the World Health Organization (WHO) 2008 classification (at Screening);
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (at the time the participant signs their first ICF);
5. Presence of FLT3-ITD activating mutation in bone marrow (allelic ratio of ≥3% FLT3-ITD/total FLT3);
6. Participant is receiving standard "7+3" induction chemotherapy regimen as specified in the protocol;
7. Adequate renal function defined as:

   a. Creatinine clearance >50 mL/min, as calculated with the modified Cockcroft Gault equation
8. Adequate hepatic function defined as:

   1. Total serum bilirubin (TBL) ≤1.5 × upper limit of normal (ULN) unless the participant has documented Gilbert's syndrome or the increase is related to increased unconjugated (indirect) bilirubin due to hemolysis;
   2. Serum alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 × ULN;
9. Serum electrolytes within normal limits: potassium, calcium (total, or corrected for serum albumin in case of hypoalbuminemia or ionized calcium) and magnesium. If outside of normal limits, participant will be eligible when electrolytes are corrected;
10. If a woman of childbearing potential, must have a negative serum pregnancy test upon entry into this study and must be willing to use highly effective birth control upon enrollment, during the treatment period and for 6 months following the last dose of investigational drug or cytarabine, whichever is later. A woman is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months);
11. If male, must be surgically sterile or willing to use highly effective birth control upon enrollment, during the treatment period, and for 6 months following the last dose of investigational drug or cytarabine, whichever is later.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL), French-American-British classification M3 or WHO classification of APL with translocation, t(15;17)(q22;q12), or breakpoint cluster region-Abelson murine leukemia viral oncogene homolog 1 (BCR-ABL) positive leukemia (ie, chronic myelogenous leukemia in blast crisis); participants who undergo diagnostic workup for APL and treatment with all-trans retinoic acid (ATRA), but who are found not to have APL, are eligible (treatment with ATRA must be discontinued before starting induction chemotherapy).
2. Diagnosis of AML secondary to prior chemotherapy or radiotherapy for other neoplasms;
3. Prior treatment for AML, except for the following allowances:

   * Leukapheresis;
   * Treatment for hyperleukocytosis with hydroxyurea;
   * Cranial radiotherapy for central nervous system (CNS) leukostasis;
   * Prophylactic intrathecal chemotherapy;
   * Growth factor/cytokine support;
4. Prior treatment with quizartinib or other FLT3-ITD inhibitors;
5. Prior treatment with any investigational drug or device within 30 days prior to Randomization (within 2 weeks for investigational or approved immunotherapy) or currently participating in other investigational procedures;
6. History of known CNS leukemia, including cerebrospinal fluid positive for AML blasts; lumbar puncture is recommended for participants with symptoms of CNS leukemia to rule out extramedullary CNS involvement;
7. History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for at least 2 years;
8. Uncontrolled or significant cardiovascular disease, including any of the following:

   * Bradycardia of less than 50 beats per minute, unless the participant has a pacemaker;
   * Fridericia's Heart Rate Correction Formula (QTcF) interval >450 msec;
   * Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
   * Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg;
   * History of clinically relevant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes);
   * History of second (Mobitz II) or third degree heart block (participants with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker);
   * History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening;
   * History of New York Heart Association Class 3 or 4 heart failure;
   * Known history of left ventricular ejection fraction (LVEF) ≤45% or less than the institutional lower limit of normal;
   * Complete left bundle branch block;
9. Active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial or antiviral therapy;
10. Known active clinically relevant liver disease (eg, active hepatitis B, or active hepatitis C);
11. Known history of human immunodeficiency virus (HIV). Participants should be tested for HIV prior to Randomization if required by local regulations or EC;
12. History of hypersensitivity to any excipients in the quizartinib/placebo tablets;
13. Females who are pregnant or breastfeeding;
14. Otherwise considered inappropriate for the study by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (244):
- United States (11):
  - University of Florida (UF) Health Shands Hospital, Gainesville, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Franciscan St. Francis Health Indianapolis, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - NY Medical College - Hudson Valley Hematology Oncology Associates, Valhalla, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - West Virginia University Hospitals, Inc., Morgantown, West Virginia
- Argentina (2):
  - Sanatorio Britanico, Rosario, Santa Fe Province
  - Sanatorio Allende, Córdoba
- Australia (4):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Townsville Hospital (TTH), Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - UCL Mont-Godinne, Yvoir
- Brazil (6):
  - Hospital Amaral Carvalho, Brasília
  - Hospital do CEPON, Brasília
  - Instituto do Cancer do Estado de São Paulo, Brasília
  - Santa Casa de Misericórdia de Porto Alegre, Brasília
  - Hospital da Cidade de Passo Fundo, Passo Fundo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment "Dr. G. Stranski" EAD, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Sofia
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital (VGH), Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (11):
  - Peking University First Hospital, Beijing
  - The General Hospital of People's Liberation Army (301 Hospital), Beijing
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai
  - West China Hospital, Sichuan University, Taiyuan
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tang Du Hospital, Fourth Military Medical University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Croatia (3):
  - Klinička Bolnica Dubrava, Zagreb
  - Klinička Bolnica Merkur, Zagreb
  - Klinički Bolnički Centar Zagreb, Zagreb
- Czechia (5):
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní Nemocnice Olomouc, Olomouc
  - Fakultní Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, Pilsen
  - Vseobecna Fakultni Nemocnice, Ustav hematologie a krevni transfuze (UHKT), Prague
- France (13):
  - Hospital A. Michallon, Grenoble
  - Centre Hospitalier de Versailles - Hôpital André Mignot, Le Chesnay
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - L'Institut Paoli - Calmettes, Marguerittes
  - Hôpital de la Conception, Marseille
  - CHRU Montpellier - Saint Eloi, Montpellier
  - Hôpital Saint-Antoine, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel - Centre de Lutte Contre le Cancer, Rouen
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Purpan, Toulouse
- Germany (15):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charité - Universitätsmedizin Berlin, Berlin
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Marien Hospital Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Halle
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Medizinische Hochschule Hannover (MHH), Hannover
  - Universitätsklinikum Münster, Heidelberg
  - Universitätsklinikum Tübingen, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - HELIOS Klinikum Wuppertal, Wuppertal
- Prince of Wales Hospital, Shatin, Hong Kong
- Hungary (6):
  - Markusovszky Egyetemi Oktatókórház, Budapest
  - Szegedi Tudományegyetem, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Központ, Pécs
  - Markusovszky Egyetemi Oktatókórház, Szombathely
- Israel (7):
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov, Tsifrin
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah University Medical Center, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (24):
  - Azienda Ospedaliera Nazionale SS.Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Sanitaria Locale 13 - Ospedale "C. e G. Mazzoni"- Ascoli Piceno, Ascoli Piceno
  - Azienda Ospedaliero - Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - IRCCS AOU San Martino - IST, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - A.O.R.N. "A. Cardarelli", Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Ospedale S. Maria delle Croci - Ravenna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale S. Eugenio, Roma
  - Policlinico Tor Vergata, Roma
  - IRCCS Ospedale San Raffaele, Roma
  - Azienda Ospedaliero-Universitaria Careggi, Roma
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Roma
  - Azienda Ospedaliera Universitaria "Federico II", Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria OO.RR. San Giovanni di Dio Ruggi d'Aragona, Salerno
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - ASST dei Sette Laghi - Ospedale di Circolo e Fondazione Macchi Varese, Varese
- Japan (29):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - University of Fukui Hospital, Yoshida, Fukui
  - Kyushu University Hospital, Higashi, Fukuoka
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Gunma University Hospital, Maebashi, Gunma
  - Chugoku Central Hospital, Fukuyama, Hiroshima
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Sendai Medical Center, Sendai, Miagi
  - Tenri Hospital, Tenri, Nara
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center, Komagome Hospital, Bunkyō-Ku, Tokyo
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Akita University Hospital, Akita
  - Aomori Prefectural Central Hospital, Aomori
  - Chiba Aoba Municipal Hospital, Chiba
  - Kameda Medical Center - Kameda General Hospital, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Gifu Municipal Hospital, Gifu
  - National Hospital Organization Kagoshima Medical Center, Kagoshima
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - Osaka City General Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - NTT Medical Center Tokyo, Tokyo
- Poland (4):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewódzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - Instytut Hematologii i Transfuzjologi, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr. 1 we Wrocławiu, Warsaw
- Portugal (5):
  - Centro Hospitalar e Universitário de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Central, EPE - Hospital Santo António dos Capuchos, Lisbon
  - Centro Hospitalar do Porto, EPE - Hospital Geral de Santo António, Porto
  - Instituto Português Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de São João, EPE - Hospital de São João, Porto
- Romania (9):
  - Institutul Regional de Oncologie Iași, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuţă" Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Spitalul Clinic Judetean de Urgenta Târgu-Mureş (4005), Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Târgu-Mureş (4008), Târgu Mureş
- Russia (9):
  - Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - Penza Regional Oncology Dispensary, Penza
  - Republican Hospital n.a.V.A. Baranov, Petrozavodsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Russian Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - Leningrad Regional Clinic and Hospital, Saint Petersburg
  - Almazov Federal North-West Medical Research Centre, Saint Petersburg
  - Saratov State Medical University named after V.I. Razumovsky, Saratov
  - Tula Regional Clinical Hospital, Tula
- Serbia (3):
  - Klinički Centar Srbije, Belgrade
  - Klinički Centar Niš, Niš
  - Klinički Centar Vojvodine, Novi Sad
- Singapore (2):
  - National University Hospital (S) Pte Ltd, Singapore
  - Singapore General Hospital, Singapore
- South Korea (18):
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SoonChunHyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Sŏwŏn
  - Ulsan University Hospital (UUH), Ulsan
- Spain (37):
  - Hospital Universitari Son Espases, Palma, Mallorca
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete - Hospital General Universitario, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Catalan Institute of Oncology (ICO), Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Complejo Hospitalario Universitario Granada, Granada
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirón Madrid, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Fundación Jiménez Díaz, Pamplona
  - Hospital Clínico Universitario "Lozano Blesa", Pamplona
  - Hospital General Universitario Morales Meseguer, Pamplona
  - Hospital Universitario Miguel Servet, Pamplona
  - Hospital Álvaro Cunqueiro, Pamplona
  - Hosp Universitario Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complexo Hospitalario Universitario de Santiago (CHUS) - Hospital Clínico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City, Niaosong District
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- Ukraine (4):
  - Cherkasy Regional Oncology Dispensary, Cherkasy
  - Poltava Regional Clinical Hospital named after M. V. Sklifosovskoho, Poltava
  - Vinnitsa Regional Clinical Hospital im. N.I. Pirogov, Vinnytsia
  - Zhitomir Regional Clinical Hospital, Zhytomyr
- Maidstone and Tunbridge Wells NHS Trust - Maidstone Hospital, Maidstone, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Levis MJ, Erba HP, Montesinos P, Kim HJ, Vrhovac R, Patkowska E, Zak P, Wang PN, Connolly Rohrbach JE PhD, Chang K, Liu L, Mostafa Kamel Y, Imadalou K, Lesegretain A, Cortes JE, Sekeres MA, Dombret H, Amadori S, Wang J, Schlenk RF, Perl AE. FLT3-ITD measurable residual disease from the QuANTUM-First trial. Blood Adv. 2025 Oct 6:bloodadvances.2025016444. doi: 10.1182/bloodadvances.2025016444. Online ahead of print. PMID 41052406
- [Derived] Schlenk RF, Montesinos P, Kim HJ, Romero-Aguilar A, Vrhovac R, Patkowska E, Zak P, Wang PN, Hanyok J, Liu L, Kamel YM, Imadalou K, Lesegretain A, Cortes J, Sekeres MA, Dombret H, Amadori S, Wang J, Perl AE, Levis MJ, Erba HP. Impact of hematopoietic cell transplantation and quizartinib in newly diagnosed patients with acute myeloid leukemia and FMS-like tyrosine kinase 3-internal tandem duplications in the QuANTUM-First trial. Haematologica. 2025 Sep 1;110(9):2024-2039. doi: 10.3324/haematol.2024.286623. Epub 2025 Mar 13. PMID 40079105
- [Derived] Erba HP, Montesinos P, Kim HJ, Patkowska E, Vrhovac R, Zak P, Wang PN, Mitov T, Hanyok J, Kamel YM, Rohrbach JEC, Liu L, Benzohra A, Lesegretain A, Cortes J, Perl AE, Sekeres MA, Dombret H, Amadori S, Wang J, Levis MJ, Schlenk RF; QuANTUM-First Study Group. Quizartinib plus chemotherapy in newly diagnosed patients with FLT3-internal-tandem-duplication-positive acute myeloid leukaemia (QuANTUM-First): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 May 13;401(10388):1571-1583. doi: 10.1016/S0140-6736(23)00464-6. Epub 2023 Apr 25. PMID 37116523
- [Derived] Cortes J, Perl AE, Dohner H, Kantarjian H, Martinelli G, Kovacsovics T, Rousselot P, Steffen B, Dombret H, Estey E, Strickland S, Altman JK, Baldus CD, Burnett A, Kramer A, Russell N, Shah NP, Smith CC, Wang ES, Ifrah N, Gammon G, Trone D, Lazzaretto D, Levis M. Quizartinib, an FLT3 inhibitor, as monotherapy in patients with relapsed or refractory acute myeloid leukaemia: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2018 Jul;19(7):889-903. doi: 10.1016/S1470-2045(18)30240-7. Epub 2018 May 31. PMID 29859851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 539 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment at 193 study sites in the following countries: Spain, Italy, Republic of Korea, Japan, China, US, France, Brazil, Germany, Russian Federation, Taiwan, Hungary, Czech Republic, Romania, Israel, Canada, Serbia, Poland, Portugal, Australia, Belgium, Bulgaria, Croatia, Ukraine, Singapore, and the UK. A total of 6 participants were randomized, but did not received treatment.
Groups:
- Quizartinib: Participants who were randomized to receive quizartinib treatment regimen.
- Placebo: Participants who were randomized to receive placebo treatment regimen.
Period: Overall Study
Arm/Group | Quizartinib | Placebo
Started | 268 | 271
Safety Analysis Set | 265 | 268
Completed | 56 | 52
Not Completed | 212 | 219
Not completed — Refractory disease | 41 | 70
Not completed — Relapse | 44 | 65
Not completed — Adverse Event | 58 | 23
Not completed — Subject decision to stop study drug | 25 | 23
Not completed — Other reasons not specified | 16 | 11
Not completed — Non-protocol-specified AML therapy | 12 | 6
Not completed — Investigator decision | 10 | 7
Not completed — Failure to meet continuation criteria | 5 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Intent-to-Treat Analysis Set.
Groups:
- Quizartinib: Participants who were randomized to receive the quizartinib treatment regimen.
- Total: Total of all reporting groups
Arm/Group | Quizartinib | Placebo | Total
Number analyzed (Participants) | 268 | 271 | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.07) | 54.3 (12.81) | 54.0 (12.93)
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 161 | 162 | 323
  ≥60 years | 107 | 109 | 216
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 150 | 294
  Male | 124 | 121 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 80 | 78 | 158
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 159 | 163 | 322
  Other | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 6 | 2 | 8
  United States | 8 | 13 | 21
  Czechia | 17 | 15 | 32
  Portugal | 3 | 6 | 9
  Russia | 13 | 6 | 19
  South Korea | 36 | 34 | 70
  China | 9 | 11 | 20
  Brazil | 7 | 8 | 15
  Poland | 3 | 8 | 11
  Bulgaria | 1 | 1 | 2
  France | 13 | 12 | 25
  Serbia | 12 | 6 | 18
  Croatia | 5 | 10 | 15
  Romania | 6 | 11 | 17
  Hungary | 4 | 5 | 9
  Japan | 16 | 13 | 29
  Ukraine | 2 | 1 | 3
  United Kingdom | 1 | 0 | 1
  Spain | 33 | 34 | 67
  Canada | 8 | 5 | 13
  Belgium | 4 | 3 | 7
  Taiwan | 12 | 17 | 29
  Italy | 31 | 29 | 60
  Israel | 5 | 9 | 14
  Australia | 3 | 5 | 8
  Germany | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Overall survival is defined as the time from randomization until death from any cause.
Time Frame: Date of randomization to the date of death due to any cause, up to approximately 3 years after enrollment
Population: Overall survival was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
months | 31.9 [21.0 to NA] — Due to insufficient number of events, an estimate of the upper limit of the confidence interval could not be determined | 15.1 [13.2 to 26.2]
Statistical Analysis 1: Comparison: Quizartinib vs Placebo; Test type: Other; p = 0.0324, Log Rank; Stratification factors include region, age, and WBC count at the time of diagnosis of AML; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.615 to 0.979]

2. Secondary Outcome: Event-free Survival in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Event-free survival (EFS) is the time from randomization to the earliest date of either refractory disease (or treatment failure [TF]), relapse, or death from any cause. Refractory disease is defined as complete remission never achieved during Induction (CR: >1000 neutrophils, >100,000 platelets, <5% blasts, and other [defined as absence of extramedullary disease [EMD], blasts with rods, and leukemic blasts]). For refractory disease, EFS event date is Day 1 (randomization). Relapse after CR is defined as ≥5% blasts, leukemic blasts, extramedullary leukemia, and presence of rods. This analysis is based on a response assessment with TF defined as not achieving response of CR, using a 42- day window from the start of the last cycle in Induction for CR evaluation.
Time Frame: Date of randomization to the date of refractory disease, relapse, or death, up to approximately 3 years after enrollment
Population: Event-free survival was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
months | 0.03 [0.03 to 0.95] | 0.71 [0.03 to 3.42]

3. Secondary Outcome: Complete Remission (CR) Rate at the End of Induction in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Complete remission (CR) rate is defined as the percentage of participants achieving CR, defined as <5% blasts, >1000 neutrophils, >100,000 platelets, and other [defined as absence of extramedullary disease [EMD], blasts with rods, and leukemic blasts], after induction
Time Frame: Approximately Cycle 1 Day 21 (Induction) to end of Induction, up to approximately 120 days (each Induction cycle is up to 60 days)
Population: Complete remission was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
Participants | 147 | 150

4. Secondary Outcome: Composite CR Rate at the End of Induction in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Composite complete remission (CRc) rate is defined as the percentage of participants whose best response is complete remission (CR), defined as <5% blasts, >1000 neutrophils, >100,000 platelets, and other [defined as absence of extramedullary disease [EMD], blasts with rods, and leukemic blasts], or CR with incomplete neutrophil or platelet recovery (CRi) at the end of first Induction cycle.
Time Frame: as for outcome 3
Population: Composite complete remission (CRc) rate was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
Participants | 192 | 176

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Occurring in ≥10% Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occur, having been absent before first dose of quizartinib or placebo, or have worsened in severity after initiating quizartinib or placebo. Adverse events collected more than 30 days after the last dose of quizartinib/placebo will not be considered TEAEs unless they are considered drug-related.
Time Frame: Date of first dose up to 30 days after last dose, up to 36 cycles following continuation (approximately 6 years 11 months, each cycle is 28 days)
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 265 | 268
Participants
  Any TEAE | 264 | 265
  Gastrointestinal disorders | 215 | 209
  Diarrhoea | 98 | 94
  Nausea | 90 | 84
  Vomiting | 65 | 53
  Stomatitis | 57 | 56
  Constipation | 56 | 69
  Abdominal pain | 46 | 38
  Dyspepsia | 30 | 23
  Abdominal pain upper | 29 | 25
  Infections and infestations | 204 | 188
  Pneumonia | 39 | 41
  Sepsis | 15 | 28
  General disorders and administration site disorders | 177 | 173
  Pyrexia | 112 | 109
  Oedema peripheral | 30 | 37
  Fatigue | 29 | 23
  Blood and lymphatic system disorders | 168 | 143
  Febrile neutropenia | 117 | 113
  Neutropenia | 54 | 27
  Thrombocytopenia | 30 | 30
  Anaemia | 29 | 19
  Metabolism and nutrition disorders | 165 | 153
  Hypokalaemia | 93 | 96
  Decreased appetite | 46 | 36
  Hypomagnesaemia | 30 | 30
  Hypophosphataemia | 27 | 24
  Hypocalcaemia | 26 | 29
  Skin and subcutaneous tissue disorders | 152 | 158
  Rash | 69 | 66
  Pruritus | 35 | 40
  Investigations | 140 | 105
  Alanine aminotransferase increased | 42 | 27
  Electrocardiogram QT prolonged | 36 | 11
  Aspartate aminotransferase increased | 28 | 19
  Neutrophil count decreased | 27 | 12
  Respiratory, thoracic, and mediastinal disorders | 123 | 115
  Cough | 50 | 44
  Epistaxis | 40 | 29
  Oropharyngeal pain | 27 | 18
  Nervous system disorders | 103 | 97
  Headache | 73 | 53
  Musculoskeletal and connective tissue disorders | 91 | 108
  Arthralgia | 29 | 35
  Back pain | 19 | 28
  Vascular disorders | 71 | 70
  Hypertension | 29 | 33
  Psychiatric disorders | 57 | 50
  Insomnia | 37 | 30

6. Secondary Outcome: Number of Participants Achieving CR With FLT3-ITD Minimal Residual Disease Negativity at the End of Induction in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Complete remission (CR) is defined as participants achieving CR defined as <5% blasts, >1000 neutrophils, >100,000 platelets, and other [defined as absence of extramedullary disease [EMD], blasts with rods, and leukemic blasts]. Minimal or measurable residual disease is the presence of a small number of leukemic cells in the bone marrow of patients with AML below the level of detection using conventional morphologic assessment.
Time Frame: Approximately Cycle 1 Day 21 (Induction phase) to end of Induction phase, up to approximately 120 days (each Induction cycle is up to 60 days)
Population: Complete remission was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
Participants | 54 | 51

7. Secondary Outcome: Number of Participants Achieving Composite CR With FLT3-ITD Minimal Residual Disease Negativity at the End of Induction in Participants With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia
Description: Composite complete remission (CRc) is defined as <5% blasts, >1000 neutrophils, >100,000 platelets, and other [defined as absence of extramedullary disease [EMD], blasts with rods, and leukemic blasts], or CR with incomplete neutrophil or platelet recovery (CRi). Minimal or measurable residual disease is the presence of a small number of leukemic cells in the bone marrow of patients with AML below the level of detection using conventional morphologic assessment.
Time Frame: as for outcome 6
Population: Composite complete remission (CRc) rate was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib | Placebo
Number analyzed (Participants) | 268 | 271
Participants | 66 | 58

8. Secondary Outcome: Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve at Steady State
Description: AUCss was assessed by population Pharmacokinetic (PK) analysis during Cycle 1 of each phase.
Time Frame: Induction Cycle 1: Day 8, predose, 2-4 hours (hr) postdose on Days 8, 15, 21; Consolidation Cycle 1: Day 6, predose, 2-4 hr postdose on Days 6, 13, 19; Continuation Cycle 1: 2-4 hr postdose, Days 1, 8, 15; Cycle 2 Days 1 and 15 (each cycle, 28 days)
Population: PK Parameters were assessed in the PK Analyses set, which includes all participants in the Intent-to-Treat Analysis Set who received at least 1 dose of quizartinib and had at least 1 PK sample assessed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Quizartinib
Number analyzed (Participants) | 259
nanogram/milliliter (ng/mL)
  Induction Period | 2680 (84.9)
  Consolidation Period: number analyzed (Participants) | 164
  Consolidation Period | 3930 (77.6)
  Continuation Period - Dose 1: number analyzed (Participants) | 115
  Continuation Period - Dose 1 | 5080 (74.7)
  Continuation Period - Dose 2: number analyzed (Participants) | 115
  Continuation Period - Dose 2 | 10200 (74.7)

9. Secondary Outcome: Pharmacokinetic Parameter Steady State, Maximum Plasma Concentration (Css,Max)
Description: Css,max was assessed by population PK analysis during Cycle 1 of each phase.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Quizartinib
Number analyzed (Participants) | 259
nanogram/milliliter (ng/mL)
  Induction Period | 140 (71.2)
  Consolidation Period: number analyzed (Participants) | 164
  Consolidation Period | 204 (63.5)
  Continuation Period - Dose 1: number analyzed (Participants) | 115
  Continuation Period - Dose 1 | 265 (59.7)
  Continuation Period - Dose 2: number analyzed (Participants) | 115
  Continuation Period - Dose 2 | 529 (59.7)

10. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Plasma Concentration Steady State (Tmax,ss)
Description: Tmax,ss was assessed by population PK analysis during Cycle 1 of each phase.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Quizartinib
Number analyzed (Participants) | 259
hours
  Induction Period | 2.68 [1.52 to 7.30]
  Consolidation Period: number analyzed (Participants) | 164
  Consolidation Period | 2.70 [1.74 to 5.95]
  Continuation Period - Dose 1: number analyzed (Participants) | 115
  Continuation Period - Dose 1 | 2.73 [1.74 to 5.95]
  Continuation Period - Dose 2: number analyzed (Participants) | 115
  Continuation Period - Dose 2 | 2.73 [1.74 to 5.95]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from date of first dose up to 30 days after last dose, up to 36 cycles following continuation phase (approximately 6 years 11 months, each cycle is 28 days).
Groups:
- Quizartinib; Placebo: Safety Analysis Set includes all subjects who received at least 1 dose of quizartinib/placebo.
Arm/Group | Quizartinib | Placebo
All-Cause Mortality (participants affected / at risk) | 130/265 | 156/268
Serious Adverse Events (participants affected / at risk) | 146/265 | 124/268
Other Adverse Events (participants affected / at risk) | 258/265 | 258/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib (N=265) | Placebo (N=268)
Febrile neutropenia (Blood and lymphatic system disorders) | 29 | 22
Neutropenia (Blood and lymphatic system disorders) | 4 | 5
Myelosuppression (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 8
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Allergic otitis externa (Ear and labyrinth disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 4 | 0
Colitis (Gastrointestinal disorders) | 3 | 3
Neutropenic colitis (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 5
Generalised oedema (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Cyst rupture (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fat necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 4 | 0
Graft versus host disease (Immune system disorders) | 1 | 2
Pneumonia (Infections and infestations) | 17 | 15
Septic shock (Infections and infestations) | 11 | 9
Sepsis (Infections and infestations) | 10 | 14
Klebsiella sepsis (Infections and infestations) | 7 | 1
Herpes zoster (Infections and infestations) | 5 | 1
Pneumonia fungal (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
COVID-19 (Infections and infestations) | 3 | 0
Bacteraemia (Infections and infestations) | 2 | 1
Pseudomonas infection (Infections and infestations) | 2 | 1
Cellulitus (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 2 | 0
Mucormycosis (Infections and infestations) | 2 | 0
Streptococcal sepsis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 3
Endocarditis (Infections and infestations) | 1 | 2
Enterococcal sepsis (Infections and infestations) | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 2
Abdominal infection (Infections and infestations) | 1 | 1
Anal infection (Infections and infestations) | 1 | 1
Aspergillus infection (Infections and infestations) | 1 | 1
BK virus infection (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hepatosplenic candidiasis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Disseminated varicella zoster virus infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Stenotrophomonas sepsis (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Systemic mycosis (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 1
Acid base balance abnormal (Investigations) | 1 | 0
Blood magnesium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Renal failure (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Quizartinib (N=265) | Placebo (N=268)
Febrile neutropenia (Blood and lymphatic system disorders) | 98 (169) | 97 (178)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (46) | 25 (37)
Anaemia (Blood and lymphatic system disorders) | 27 (39) | 18 (35)
Neutropenia (Blood and lymphatic system disorders) | 53 (130) | 22 (29)
Dry eye (Eye disorders) | 22 (22) | 13 (17)
Diarrhoea (Gastrointestinal disorders) | 97 (146) | 94 (133)
Nausea (Gastrointestinal disorders) | 91 (168) | 84 (141)
Vomiting (Gastrointestinal disorders) | 63 (88) | 51 (76)
Stomatitis (Gastrointestinal disorders) | 56 (70) | 55 (66)
Abdominal pain (Gastrointestinal disorders) | 46 (59) | 38 (52)
Constipation (Gastrointestinal disorders) | 57 (77) | 69 (91)
Dyspepsia (Gastrointestinal disorders) | 29 (37) | 22 (27)
Hemorrhoids (Gastrointestinal disorders) | 26 (30) | 20 (24)
Abdominal pain upper (Gastrointestinal disorders) | 29 (36) | 25 (30)
Gingival bleeding (Gastrointestinal disorders) | 14 (15) | 13 (18)
Pyrexia (General disorders) | 113 (203) | 106 (224)
Oedema peripheral (General disorders) | 30 (36) | 37 (40)
Fatigue (General disorders) | 31 (44) | 23 (35)
Asthenia (General disorders) | 15 (19) | 20 (29)
Chills (General disorders) | 8 (9) | 14 (19)
Pneumonia (Infections and infestations) | 25 (29) | 27 (30)
Upper respiratory tract infection (Infections and infestations) | 20 (38) | 15 (22)
Conjunctivitis (Infections and infestations) | 16 (19) | 8 (10)
Bacteraemia (Infections and infestations) | 14 (19) | 5 (5)
Sepsis (Infections and infestations) | 5 (5) | 14 (14)
Folliculitis (Infections and infestations) | 14 (19) | 4 (5)
Oral herpes (Infections and infestations) | 17 (18) | 11 (14)
Transfusion reaction (Injury, poisoning and procedural complications) | 11 (14) | 19 (30)
Electrocardiogram QT prolonged (Investigations) | 35 (70) | 11 (12)
Alanine aminotransferase increased (Investigations) | 43 (64) | 26 (43)
Gamma-glutamyltransferase increased (Investigations) | 23 (31) | 25 (33)
Aspartate aminotransferase increased (Investigations) | 29 (41) | 19 (30)
Neutrophil count decreased (Investigations) | 24 (73) | 12 (27)
Platelet count decreased (Investigations) | 18 (34) | 7 (17)
Blood bilirubin increased (Investigations) | 15 (21) | 13 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 93 (148) | 96 (162)
Decreased appetite (Metabolism and nutrition disorders) | 46 (71) | 36 (44)
Hypocalcaemia (Metabolism and nutrition disorders) | 25 (36) | 29 (39)
Hypophosphataemia (Metabolism and nutrition disorders) | 27 (42) | 24 (32)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 23 (28) | 23 (31)
Hypomagnesaemia (Metabolism and nutrition disorders) | 30 (44) | 30 (45)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (12) | 15 (20)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (14) | 14 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (37) | 35 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (25) | 27 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (25) | 21 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (18) | 17 (19)
Headache (Nervous system disorders) | 73 (120) | 54 (101)
Dizziness (Nervous system disorders) | 17 (18) | 20 (22)
Insomnia (Psychiatric disorders) | 38 (46) | 30 (36)
Anxiety (Psychiatric disorders) | 15 (18) | 12 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 (45) | 29/265 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 49 (56) | 44 (50)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (35) | 18 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 20 (25)
Rash (Skin and subcutaneous tissue disorders) | 69 (100) | 66 (102)
Pruritus (Skin and subcutaneous tissue disorders) | 35 (49) | 40 (48)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 18 (21) | 14 (15)
Urticaria (Skin and subcutaneous tissue disorders) | 17 (23) | 11 (14)
Hypertension (Vascular disorders) | 30 (35) | 33 (40)
Hypotension (Vascular disorders) | 23 (27) | 17 (21)
Nasopharyngitis (Infections and infestations) | 14 (20) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02668653/Prot_SAP_000.pdf